CLINICAL TRIAL: NCT01056406
Title: Nutrition Intervention for the Promotion of Healthy Weight Gain During Pregnancy: The Revere Pregnancy Weight Management Study
Brief Title: Nutrition Intervention for the Promotion of Healthy Weight Gain During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alessandra Peccei, MD, Alessandra Peccei, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-P-002171/1; MGH
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Pregnancy; Overweight; Obesity
Keywords: Pregnancy; Overweight; Obese; Nutrition intervention
MeSH Terms: conditions — Overweight; Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Overweight and obese pregnant women who are randomly assigned to the control group will receive the current standard of optimal care in addition to 1 nutrition education session with the study nutritionist (a registered dietitian) at 6-16 weeks gestation.
- Nutrition Education Group (Experimental): Overweight and obese pregnant women randomly assigned to the nutrition education group, in addition to the current standard of optimal care, will receive twice monthly interaction with the study nutritionist (a registered dietitian) from 6-16 weeks gestation through 6 months postpartum.
  Interventions: Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: Nutrition Education — Twice monthly interaction with study nutritionist (a registered dietitian) in the form of face-to-face individual nutrition counseling sessions, telephone and electronic follow-ups, option to attend group nutrition and group exercise classes.
  Arms: Nutrition Education Group

SUMMARY:
The purpose of this study is to determine if twice monthly interaction with a registered dietitian from 6-16 weeks gestation through 6 months postpartum will help women who are overweight or obese gain weight during pregnancy closer to the Institute of Medicine (IOM)guidelines and lose weight more effectively within the 6 month postpartum period than those who do not receive twice monthly interaction with a registered dietitian during this period.

Overweight/obesity can lead to a number of adverse pregnancy, delivery and birth outcomes, including increased risk of hypertension, eclampsia, and diabetes during pregnancy, miscarriage, premature delivery, birth injuries, neural tube defects, and prenatal death. More than half of women of childbearing age are overweight or are obese. Women of color and low-income women are affected disproportionately.

Unfortunately, women know little, if anything, about the impact of overweight and obesity on pregnancy and health care providers are unsure how to effectively address the problem with their patients.

A limited number of programs have tested ways to effectively address weight gain management during pregnancy. None have been successful in addressing weight gain in women who are obese or overweight at the start of pregnancy. The 2-year Revere Health Center Pregnancy Weight Management Study will test the feasibility and efficacy of providing pregnant women who are overweight or obese with regular access to a registered dietitian during and after pregnancy to help achieve total weight gain closer to recommended guidelines and to ensure the best outcomes for the mother and her newborn.

DETAILED DESCRIPTION:
The Revere Pregnancy and Weight Management Study has been designed to test the hypothesis that women with a BMI > 25 and < 40 who receive information about the risks of excessive weight gain during pregnancy and bimonthly interventions from a registered dietitian from the beginning of their pregnancy (6-16 weeks gestation) through 6 months postpartum, will achieve total weight gain closer to IOM (Institute of Medicine) guidelines and will have fewer complications as compared to women who only receive information about the risks of excessive weight gain (i.e. Current standard of optimal care). In addition, we hope to find that women who participate in the program will increase physical activity and show improvement in overall nutritious food choices as will be measured by the results of a nutrition and physical activity questionnaire completed by all participants at 3 points during the study.

This study will be managed completely by a registered dietitian who has experience working with pregnant women. The dietitian will have direct access to the participants' primary clinicians for consultation throughout the course of the study.

All patients, regardless of whether in the control or intervention group, will receive the optimal standard of prenatal and postpartum care and any additional care needed to ensure the best outcomes for the mother and newborn.

Everyone in the study will meet with the dietitian who works at the Revere Health Center at least one time. During the initial visit, participants will receive information about healthy eating and exercise during pregnancy. Women will also receive information about risks to mother and baby related to excessive weight gain during pregnancy for overweight and obese women.

Women in the control group will have no further interaction with the study dietitian.

Women in the intervention group will meet with the dietitian at least twice per month. The contact with the dietitian may include face-to-face individual counseling, telephone or e-mail follow-up, group classes or group activities.

Data that will be collected and analyzed will include:

* Demographic information
* Medical and Pregnancy History
* Pregnancy, labor, and delivery complications to mother and baby
* Birth record
* Weight change during pregnancy and after delivery
* Changes in physical activity and food choices

Through bimonthly contact with the dietitian, women will learn about healthier eating habits and exercise while monitoring weight gain to help adhere to IOM guidelines. We hope to see improved pregnancy, labor, and delivery outcomes for mothers and babies and help women achieve postpartum weight loss. We intend to foster an increased interest and knowledge about nutrition that will carry over to healthier food choices to share with their families and with other women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ages 18 to 49 with a BMI >25 and <40 at the first prenatal visit
* Women < 16 weeks gestation
* Both women who have and have not received previous nutritional counseling
* Both women who have and have not dieted in the past
* Women with a documented medical history or who report a history of disordered eating including over eating, night eating, or binge eating without a diagnosis listed in the "exclusion criteria" will not be excluded

Exclusion Criteria:

* Pregnant women over age 49
* Pregnant women ages 18 to 49 with a BMI <25 or > 40 at their first prenatal visit
* Women > 16 weeks gestation
* Women pregnant with multiples
* Diabetes prior to pregnancy
* Women with a documented medical history of an eating disorder including anorexia nervosa, bulimia nervosa, anorexia athletica, and orthorexia will be excluded

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2009-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percent of total weight gained during pregnancy compared to current Institute of Medicine Guidelines. | Weight at first prenatal care appointment. Weight at last obstetrical appointment prior to delivery.

SECONDARY OUTCOMES:
Overall improvement of the intake of nutritious foods as quantified by a written nutrition and exercise questionnaire. | Enrollment, 6 weeks postpartum, 6 months postpartum
Prevalence of complications, specifically: -hypertension and eclampsia, -gestational diabetes, -caesarian delivery, -macrosomia -admission to neonatal intensive care unit (NICU) | Throughout study participation
Initiation of breastfeeding | 6 weeks postpartum
Postpartum weight reduction in comparison to pre-pregnancy baseline weight (BMI) | 6 month postpartum
Maintenance of improvements in overall intake of nutritious foods as quantified by the nutrition and exercise questionnaire | 6 weeks post partum, 6 months postpartum
Maintenance of improvements in physical activity as quantified by the nutrition and exercise questionnaire | 6 weeks postpartum, 6 months postpartum
Maintenance of breastfeeding | 6 weeks postpartum, 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Peccei, MD, Study Director — Partners HealthCare System at Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital HealthCare Center Revere, Revere, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
in process

REFERENCES:
- [Derived] Peccei A, Blake-Lamb T, Rahilly D, Hatoum I, Bryant A. Intensive Prenatal Nutrition Counseling in a Community Health Setting: A Randomized Controlled Trial. Obstet Gynecol. 2017 Aug;130(2):423-432. doi: 10.1097/AOG.0000000000002134. PMID 28697099